CLINICAL TRIAL: NCT03751319
Title: Geriatric Assessment and Intervention for Older Patients With Frailty in the Emergency Department. Randomized Controlled Trial
Brief Title: Geriatric Assessment and Intervention for Older Patients With Frailty in the Emergency Department
Acronym: GAOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: City of Espoo (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Janne Alakare, Senior physician in Emergency Medicine, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TYH2018304; HUS1171/2018 (Other: Helsinki University Hospital)
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Frail Elderly Syndrome; Patient Admission; Hospital Readmission; Length of Stay; Fall; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Emergency Care + CGA (Active Comparator): Standard Care is provided for the acute condition as usual by the ED personnel. Besides the standard care provided by ED personnel, patients are systemically screened and assessed by physician trained for geriatrics or geriatric emergency medicine. Geriatric multi-discipline treatment plan and recommendations are given if suitable for the case.
  Interventions: Other: CGA
- Standard Emergency Care (No Intervention): Standard Care is provided for the acute condition as usual by the ED personnel.

INTERVENTIONS:
Other: CGA — Comprehensive Geriatric Assessment
  Arms: Standard Emergency Care + CGA

SUMMARY:
Comprehensive Geriatric Assessment (CGA) is an established approach for better detection of frailty-related problems and includes individualized treatment plan with multi-discipline supportive and treating measures for the older frailty patients. However, there is limited evidence of feasibility and efficacy of the CGA when provided in the emergency department setting.

In the GAOPS-study the efficacy of the CGA in emergency department setting will be studied by randomized controlled study protocol. We aim to study if the CGA provided in the ED is feasible, safe and efficient method when added with standard emergency care for older frail patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of minimum 75 years
* "Clinical Frailty Scale" minimum 4 estimated at the arrival to the ED by nurse

Exclusion Criteria:

* Non-resident of the counties (City of Espoo, Kirkkonummi, Kauniainen) of the hospital district.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 432 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Cumulated Length of Stay | Day 365
  Cumulated stay (days) in hospital wards (university hospital and community hospital) including all admissions during the follow-up.

SECONDARY OUTCOMES:
Admissions | Day 30, Day 365
  Number of admissions to the hospital wards (university hospital and community hospital) during the follow-up.
Admission rate | Day 0
  Proportion of admitted patients (university hospital or community hospital ward) from the index ED-visits.
Readmissions in the ED | Hour 72, Day 30, Day 365
  Re-visits to the ED after the index-visit.
Living at home | Day 365
  Proportion of the patients living at home.
Quality of Life | Day 0, Day 365
  Change of the quality of life during one year follow-up using the standardized questionnaire EuroQol EQ-5D-5L. Measured value is the index value defined by the EuroQol group.

OTHER OUTCOMES:
Length-of-Stay in the ED | Day 0
  Length-of-Stay (h) of the index-visit in the ED
Length-of-Stay in the ward | Day 365
  Length-of-Stay (d) in the hospital ward of admitted patients from the index-visit in the ED
Mortality | Day 365
  Mortality during the one-year follow-up.
Falls | Day 365
  Number of falls which result in new ED visit during the one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Veli-Pekka Harjola, Study Director — Department of Emergency Medicine and Services, Helsinki University Hospital; Janne Alakare, MD, Principal Investigator — Department of Emergency Medicine and Services, Helsinki University Hospital
Locations (1):
- Helsinki University Hospital, Jorvi ED, Espoo, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alakare J, Kemp K, Strandberg T, Castren M, Jakovljevic D, Tolonen J, Harjola VP. Systematic geriatric assessment for older patients with frailty in the emergency department: a randomised controlled trial. BMC Geriatr. 2021 Jul 2;21(1):408. doi: 10.1186/s12877-021-02351-2. PMID 34215193
- See also: Alakare, J., Kemp, K., Strandberg, T. et al. Systematic geriatric assessment for older patients with frailty in the emergency department: a randomised controlled trial. BMC Geriatr 21, 408 (2021). https://doi.org/10.1186/s12877-021-02351-2 — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-021-02351-2